CLINICAL TRIAL: NCT06447779
Title: A Multicenter, Randomized, Double-Blinded, Placebo-Controlled Phase III Clinical Trial to Evaluate Efficacy, Safety and Immunogenicity of Recombinant Zoster Vaccine (CHO Cell) in Adults Aged 40 Years and Above
Brief Title: Efficacy, Safety and Immunogenicity Study of Recombinant Zoster Vaccine(CHO Cell) in Adults Aged 40 Years and Older
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: MAXVAX Biotechnology Limited Liability Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MKKCT-100-003
Record Dates: First submitted 2024-06-02; First posted 2024-06-07 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-05

CONDITIONS: Herpes Zoster
MeSH Terms: conditions — Herpes Zoster

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Vaccine Group (Experimental): Subjects will receive Recombinant Zoster Vaccine (CHO cell) according to a 0, 2-month schedule
  Interventions: Biological: Recombinant Zoster Vaccine (CHO Cell)
- Placebo Group (Placebo Comparator): Subjects will receive NaCl solution placebo according to a 0, 2-month schedule
  Interventions: Biological: NaCl solution Placebo

INTERVENTIONS:
Biological: Recombinant Zoster Vaccine (CHO Cell) — 0.5 mL per dose, containing a total of 50 µg recombinant varicella zoster virus glycoprotein E, adjuvanted with MA105.
  Intramuscular injection
  Arms: Vaccine Group
Biological: NaCl solution Placebo — 0.5 mL per dose, containing 4.5 mg sodium chloride. Intramuscular injection
  Arms: Placebo Group

SUMMARY:
The purpose of the sutdy is to evaluate efficacy, safety and immunogenicity of Recombinant Zoster Vaccine (CHO Cell) with 2 doses at 2-month interval in adults aged 40 years and older.

DETAILED DESCRIPTION:
A total of 25000 adults aged 40 years and older will be enrolled, stratified into 40-49, 50-59, 60-69 and ≥70 years of age. All subjects will randomly receive investigational vaccine or placebo at a ratio of 1:1. Efficacy and safety will be assessed in all subjects, while immunogenicity will be assessed in a subset of 1250 subjests in a selected trial site.

ELIGIBILITY:
Inclusion Criteria:

1. A male or famale permanent resident aged 40 years and older at enrollment, with valid identity;
2. Subjects voluntarily agree to participate in the study and signed an informed consent;
3. Be able to understand clinical trials, participate in all scheduled visits and comply with the protocol requirements(e.g. completion of the diary cards/questionnaires, return for follow-up visits, have regular contact to allow evaluation during the study);
4. Women of childbearing potential plan to aviod pregnancy and are willing to use effcetive contraception(e.g. oral contraceptive pills, injectable progestogen, percutaneous contraceptive patches, implants of levonorgestrel, intrauterine device, female and male sterilization or abstinence) within 12 months after the last vaccination, and the uses of the rhythm method alone, withdrawal alone, and emergency contraception, are not acceptable.

Exclusion Criteria:

1. Axillary temperature>37.0℃;
2. Current or history of herpes zoster;
3. Previous vaccination against varicella or herpes zoster (either registered product or participation in a previous vaccine study);
4. Pregnant (urine pregnancy test was positive) or lactating female;
5. Receipt of live vaccine within 28 days, or any other vaccine within 14 days prior to vaccination;
6. Receipt of immunoglobulin or intravenous immunoglobulin during 3 months before vaccination to 1 month post the last vaccination;
7. Acute diseases or acute exacerbation of chronic disease within 3 days before vaccination;
8. Receipt of antipyretic, analgesic and allergy drugs within 3 days before vaccination, except enteric-coated aspirin for cardiovascular diseases prevention;
9. A known allergy to any components of the study vaccine, or history of severe allergy (e.g. Anaphylactic shock, allergic laryngeal edema, anaphylactoid purpura, thrombocytopenic purpura, Arthus reaction, severe urticaria) to any previous vaccination;
10. Allergy to aminoglycoside antibiotics;
11. History of convulsions, epilepsy, encephalopathy (e.g. congenital brain dysplasia, brain trauma, brain tumor, cerebral hemorrhage, cerebral infarction, brain infection disease, nerve tissue damage caused by chemical drug poisoning), mental illness and family history, and other serious neurological diseases;
12. Asplenia or functional asplenia, or splenectomy caused by any condition;
13. Primary or secondary impairment of immune function, diagnosed congenital or acquired immunodeficiency, human immunodeficiency virus (HIV) infection, lymphoma, leukemia, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease or other autoimmune diseases;
14. Receipt of immunosuppressive therapy (e.g. long-term use of systemic glucocorticoid ≥14 days, dose ≥2mg/kg/day or ≥20mg/day prednisone or equivalent dose) during 6 months before vaccination to 1 minth post the last vaccination, but inhaled, nasal spray, intra-articular, eyedrops, ointment and other topical steroids are acceptable;
15. Receipt of long-acting immune-modifying drugs (e.g. Infliximab) within 6 months before vaccination or during the study period;
16. Severe chronic disease, including but not limited to, severe cardiovascular disease(e.g. Pulmonary heart disease, Pulmonary Edema), severe liver or kidney disease, or diabetes with complication;
17. History of thrombocytopenia or other coagulation disorders, which may cause intramuscular injection contraindications;
18. Abnormal and uncontrlled blood pressure during physical examination before vaccination (for subjects aged 40-59: systolic pressure ≥ 140 mmHg and/or diastolic pressure ≥ 90 mmHg; for subjects aged ≥60, systolic pressure ≥ 150 mmHg and/or diastolic pressure ≥ 100 mmHg);
19. History of drug abuse (narcotic drugs, psychotropic drugs);
20. Current skin infections, in the opinion of the investigator, might interfere with the efficacy evaluation;
21. Current or history of malignant tumors, except papillary thyroid carcinoma;
22. Receipt of investigational products (drugs or vaccines) within 6 months before vaccination;
23. Planned participation in another clinical study during the study period;
24. Any condition that, in the opinion the investigator, may affect the safety of the subject or the evaluation of the study results.

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25000 (Estimated)
Dates: Start 2024-07-13 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Incidence of confirmed Herpes Zoster(HZ) Cases per person years in subjects aged 40 years and older | 30 days after the last vaccination
  A suspected case of HZ was confirmed either: by Polymerase Chain Reaction (PCR) or by the Endpoint Adjudication Committee (EAC), consisting of physicians with HZ expertise.

SECONDARY OUTCOMES:
Incidence of confirmed Herpes Zoster(HZ) Cases per person years in different age group. | 30 days after the last vaccination
  All subjects will be stratified into 40-49 years, 50-59 years, 60-69 years and ≥70 years of age.
Incidence of any and severe Postherpetic Neuralgia (PHN) cases per person years in subjects aged 40 years and older, 40-49years , 50-59 years , 60-69 years and ≥70 years , with confirmed HZ. | 30 days after the last vaccination
  PHN of any severity was defined as 0 and greater on the Zoster Brief Pain Inventory(ZBPI) questionnaire, while severe PHN rated as 3 and greater on the ZBPI questionnaire.
Geometric Mean Concentration(GMC) of anti-gE antibody and anti-VZV antibody in immunogenicity subset | At 1, 12, 24 and 36 months after the last vaccination
  Measured by ELISA
Seropositivity rate of anti-gE antibody and anti-VZV antibody in immunogenicity subset | At 1, 12, 24 and 36 months after the last vaccination
  The seropositivity rate is defined as the percentage of subjects whose antibody concentration is greater than or equal to the cut-off value.
Seroresponse rate of anti-gE antibody and anti-VZV antibody in immunogenicity subset | 30 days after the last vaccination
  The seroresponse rate is defined as the percentage of subjects who have at least a: 4-fold increase in the antibody concentration as compared to the pre vaccination antibody concentration, for subjects who are seropositive at baseline, OR, 4-fold increase in the antibody concentration as compared to the antibody concentration cut-off value for seropositivity, for subjects who are seronegative at baseline.
Geometric Mean Fold Rise (GMFR) of anti-gE antibody and anti-VZV antibody in immunogenicity subset | At 1, 12, 24 and 36 months after the last vaccination
  The antibody concentration at evaluted time points compared with that at baseline.
Four-fold increase rate of anti-gE antibody and anti-VZV antibody in immunogenicity subset | 30 days after the last vaccination
  The antibody concentration 30 days after the last vaccination compared with that at baseline.
Cell-Mediated Immunity (CMI) response | 30 days after the last vaccination
  CMI response is defined as the frequency of CD4+ T cells producing at least 2 activation markers (IFN-γ, IL-2, TNF-α and/or CD40L) upon in vitro stimulation by gE peptide pools.
Vaccine Response Rate (VRR) | 30 days after the last vaccination
  VRR is defined as the percentage of subjects with at least a 2-fold increase as compared to the Cut-off, for subjects with pre-vaccination T-cell frequencies<Cut-off, OR, at least a 2-fold increase as compared to pre-vaccination T-cell frequencies for subjects with pre-vaccination T-cell frequencies ≥Cut-off.
Number of Participants With solicited local symptoms | Within 7 days after each vaccination
  Assessed solicited local symptoms were pain, Induration, swelling, redness, pruritus, rash, and cellulitis.
Number of Participants With solicited general symptoms. | Within 7 days after each dose
  Assessed solicited general symptoms were fever [defined as axillary equal to or above 37.3 degrees Celsius (°C)], diarrhoea, anorexia, vomiting, nausea, abdominal pain, myalgia, arthralgia, headache, syncope, new convulsions, cough, pruritus (non-vaccination site), skin and mucous membrane abnormalities, acute allergic reactions, fatigue, pain (non-vaccination site), chills.
Number of Participants With unsolicited adverse events | During 30 days after each vaccination
  An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms.
Number of Participants With Serious Adverse Events | From the day of first vaccination up to 12 months after last vaccination
  Serious adverse events (SAEs) assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization, result in disability/incapacity or is a congenital anomaly/birth defect in the offspring of a study subject.
Number of Participants With potential Immune Mediated Disorders | From the day of first vaccination up to 12 months after last vaccination
  pIMDs are a subset of Adverse Events of Specific Interest (AESIs) that include autoimmune diseases and other inflammatory and/or neurologic disorders of interest which may or may not have an autoimmune aetiology.

CONTACTS AND LOCATIONS:
Overall Officials: Wang Yanxia, Principal Investigator — Henan Center for Disease Control and Prevention
Locations (4):
- China (4):
  - Hebei Provincial Center for Disease Control and Prevention, Shijiazhuang, Hebei
  - Henan Center for Diseases Control and Prevention, Zhengzhou, Henan
  - Hubei Provincial Center for Disease Control and Prevention, Wuhan, Hubei
  - Yunnan Center For Disease Control and Prevention, Kunming, Yunnan

IPD SHARING:
Plan to Share IPD: No